CLINICAL TRIAL: NCT03575507
Title: Safety and Patient Satisfaction With Noninvasive Repetitive Pulse Magnetic Stimulation (rPMS) for Aesthetic Improvements of Buttocks
Brief Title: Non-invasive Improvement of Buttocks With Magnetic Device
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: It wasn't possible to recruit the desired number of patients.
Sponsor: BTL Industries Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTL-Buttocks_002
Record Dates: First submitted 2018-06-19; First posted 2018-07-02 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Muscle Tightness
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Treatment Group (Experimental): Treatment with the investigational device BTL EMSCULPT.
  Interventions: Device: Treatment with BTL EMSCULPT device.

INTERVENTIONS:
Device: Treatment with BTL EMSCULPT device. — The treatment administration phase will consist of four (4) treatments, delivered twice a week. The applicator will be applied over the buttock area. Visible contractions will be induced by the device.

SUMMARY:
This study will evaluate the clinical safety and patient satisfaction with the high power magnet system for the aesthetic improvement of buttocks. The study is a prospective multi-center open-label single-arm study. The subjects will be enrolled and assigned into a single study group. Subjects will be required to complete four (4) treatment visits and three follow-up visits - 1 month, 3 months and 12 months after the final treatment. Study will be conducted at several study sites.

At the baseline visit, subject's weight will be recorded.

The treatment administration phase will consist of four (4) treatments, delivered twice a week. The applicator will be applied over the gluteal area. Visible contractions will be induced by the device.

At the last therapy visit, the subject's weight will be recorded. In addition, subjects will receive Subject Satisfaction Questionnaire to fill in.

Safety measures will include documentation of adverse events (AE) including subject's experience of pain or discomfort after the procedure. Following each treatment administration and at the follow-up visits, subjects will be checked for immediate post-procedure adverse event assessment.

Post-procedure evaluation (follow-up visits) will be conducted 1 month, 3 months and 12 months after the final treatment. A weight measure will be conducted. Also, subject's satisfaction will be noted.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily signed informed consent form
* BMI ≤ 30 kg/m2
* Women of child-bearing potential are required to use birth control measures during the whole duration of the study
* Subjects willing and able to abstain from partaking in any treatments other than the study procedure to promote body contouring during study participation
* Subjects willing and able to maintain his/her regular (pre-procedure) diet and exercise regimen without effecting significant change in either direction during study participation

Exclusion Criteria:

* Cardiac pacemakers
* Electronic implants
* Pulmonary insufficiency
* Metal implants
* Drug pumps
* Haemorrhagic conditions
* Anticoagulation therapy
* Heart disorders
* Malignant tumor
* Fever
* Pregnancy
* Breastfeeding
* Following recent surgical procedures when muscle contraction may disrupt the healing process
* Application over menstruating uterus
* Application over areas of the skin which lack normal sensation
* Scars, open lesions and wounds at the treatment area
* Unrepaired abdominal hernia

Min Age: 22 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2017-06-01 (Estimated); Primary Completion 2018-09-30 (Estimated); Study Completion 2020-05-20 (Actual)

PRIMARY OUTCOMES:
Patient's satisfaction with study treatment for non-invasive aesthetic improvement of buttocks. | 18 months
  Subject's satisfaction with the therapy results evaluated through the Subject Satisfaction Questionnaire.
  The 5-point Likert scale Subject Satisfaction Questionnaire will be used for an analysis of the subject's opinion of the therapy results. Subjects will be evaluating agreement with three different statements (concerning satisfaction with therapy results and appearance of abdominal area after therapy) by choosing an answer on a scale between 1 (Strongly disagree) and 5 (Strongly agree). Minimally 80% of the treated subjects should report the agreement with all three statements given in the questionnaire (answers "Agree" and "Strongly agree") in order to claim subject's satisfaction with the therapy outcome.

SECONDARY OUTCOMES:
Determining side effects and adverse events (AE) associated with the treatment of the gluteal area. | 18 months
  The occurrence of adverse events throughout the whole study.

CONTACTS AND LOCATIONS:
Locations (2):
- Dr. Mariano Busso Aesthetic Dermatology, Miami, Florida, United States
- Aesthe Clinic, Sofia, Bulgaria

IPD SHARING:
Plan to Share IPD: No